## Official title: Client/Parent Consent Form for the "Improving Effective Mental Health Care for LGBT Clients" project

NCT number: U48DP006382

**Document date: 11/03/2020** 



Institutional Review Board
1204 Marie Mount Hall ● 7814 Regents Drive ● College Park, MD 20742 ● 301-405-4212 ● <u>irb@umd.edu</u>

## **CLIENT/PARENT CONSENT TO PARTICIPATE**

| Project Title | UMD-PRC Core Research Trial |
|---|---|
| Purpose of the Study | This research is being conducted by <b>Dr. Bradley Boekeloo</b> at the University of Maryland, College Park. We are inviting you to participate in this research project because you are 16 years or older and have been invited by your behavioral healthcare provider to participate. The purpose of this research project is to evaluate a cultural competence training program for mental healthcare providers. In this study, you will be asked to rate your satisfaction with the services you received in your last visit with that provider. |
| Procedures | The procedures involve: 1) Filling out an on-line survey that is intended to assess the behavioral health services that you have received. It asks about your demographics such as age, educational level, gender, gender identity, race/ethnicity, sexual orientation, etc., your background such as how many times you have seen your mental health provider and for what reason, as well as how you rate your experience with your provider. This survey is expected to take about 15 minutes to complete. |
| | 2) Depending on your survey responses, you may also be asked to participate in an audio-recorded on-line in-depth interview with a researcher about what you think about your mental healthcare services. This in-depth interview is expected to take about one hour to complete. If the client is 16-17 years old, they will be sent an email directly to ask if they will participate in this on-line in-depth interview. |
| Potential Risks<br>and<br>Discomforts | We anticipate minimal risk from participating in the study. You may be uncomfortable rating your provider. If you are chosen for an indepth interview, you may be uncomfortable talking with the researchers about your provider. You may also be concerned about your provider if you have negative things to say about your interaction with them. Your individual responses to study questions will not be shared with your mental health provider, their employer, or your health organization. You may skip any question you do not wish to |

| | answer. |
|---|---|
| Potential<br>Benefits | There are no direct benefits from participating in this study. However, indirect benefits include a better understanding of how to train and assess behavioral healthcare providers' in regard to their competence regarding sexuality and gender identity. |
| Confidentiality | The researchers will be collecting information from many behavioral healthcare clients and make every effort to keep all of your research information confidential from behavioral healthcare providers, their employers, or anyone else. Researchers will: Remove all names, emails, phone numbers from the dataset within 24 hours and replace this information with unique study |
| | <ul> <li>identification numbers. This information allows the researchers to match information with the provider and the organization for study purposes.</li> <li>Only share research information in reports that summarize all the information from all project participants rather than just from one person.</li> </ul> |
| | <ul> <li>Keep all information that you provide on-line in a survey stored in the University of Maryland confidential Qualtrics Survey Database Management System.</li> <li>Keep all information in audio-records of in-depth interviews in the University of Maryland Prevention Research Center password-protected computer files.</li> <li>Only access research information for research purposes under the supervision of Dr. Boekeloo.</li> </ul> |
| | Your information may be shared with representatives of the University of Maryland, College Park or governmental authorities if you or someone else is in danger or if we are required to do so by law. |
| Medical | The University of Maryland does not provide any medical, |
| Treatment | hospitalization or other insurance for participants in this research study, nor will the University of Maryland provide any medical treatment or compensation for any injury sustained as a result of participation in this research study, except as required by law. |
| Compensation | You will receive a \$20 gift card for on-line survey completion. If you are chosen for an on-line in-depth interview, you will receive a \$30 gift card for on-line in-depth interview completion. As you will not earn over \$100, only your name and address will be collected to |
| | receive compensation. |
| Right to<br>Withdraw and | Your participation in this research is completely voluntary. You may choose not to take part at all. If you decide to participate in this |

| Questions | research, you may stop participating at any time. If you decide not to participate in this study or if you stop participating at any time, you will not be penalized or lose any benefits to which you otherwise qualify. Your decision to participate or not will not affect your relationship with the mental health provider or the mental health services organization in any way. If you decide to stop taking part in the study, if you have questions, concerns, or complaints, or if you need to report an injury related to the research, please contact the investigator: Dr. Bradley Boekeloo 1142 Valley Drive College Park, MD 20742 boekeloo@umd.edu |
|---|---|
| | 301-405-4008 |
| Participant<br>Rights | If you have questions about your rights as a research participant or wish to report a research-related injury, please contact: |
| | University of Maryland College Park<br>Institutional Review Board Office<br>1204 Marie Mount Hall<br>College Park, Maryland, 20742<br>E-mail: <u>irb@umd.edu</u><br>Telephone: 301-405-0678 |
| | For more information regarding participant rights, please visit:<br>https://research.umd.edu/irb-research-participants |
| | This research has been reviewed according to the University of Maryland, College Park IRB procedures for research involving human subjects. |
| Statement of | Your signature indicates that you are at least 18 years of age. If you |
| Consent | are 16 or 17 years old, your parent/guardian must also sign this |
| | form for you to participate in this research. |
| | Your signature indicates that you have read this consent form or have had it read to you; your questions have been answered to you satisfaction and you voluntarily agree to participate in this research study. You will receive a copy of this signed consent form. If you agree to participate, please sign your name below. |
| | ii you agree to participate, please sign your name below. |
| Age of | AGE OF PARTICIPANT |

| Contact information for Participant | Email address: | Phone number: |
|---|---|---|
| Signature and Date | NAME OF PARTICIPANT [Please Print] SIGNATURE OF PARTICIPANT NAME OF PARENT (IF PARTICIPANT IS LESS THAN 18 YEARS OLD) [Please Print] SIGNATURE OF PARENT (IF PARTICIPANT IS LESS THAN 18 YEARS OLD) | |
| | DATE | |